CLINICAL TRIAL: NCT01454258
Title: Indication for Intraoperative Volume Therapy
Acronym: INDIZ_IV_I
Status: Completed | Type: Observational
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Principal Investigator, Professor Kai Zacharowski, M.D., Ph.D., FRCA, Director, Johann Wolfgang Goethe University Hospital
Other Study IDs: INDIZ IV I
Record Dates: First submitted 2011-10-14; First posted 2011-10-18 (Estimated); Results first posted 2015-12-07 (Estimated); Last update posted 2017-09-14 (Actual); Status verified 2017-08

CONDITIONS: Patients Undergoing Any Kind of Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

SUMMARY:
This study evaluates which substitution solutions are used in daily clincal practice in various teaching hospitals in a specific district (Frankfurt/Rhine-Main Metropolitan Region). Furthermore the indication for usage of these solutions is investigated.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing surgery receiving at least one bag of cristalloid or colloid solution

Exclusion Criteria:

* decline of participation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients of participating hospitals that will undergo surgery and receive intravenous fluid or volume treatment(cristalloid or colloid) will be included.
  Participating hospitals are the university teaching hospitals of the Goethe University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 10100 (Actual)
Dates: Start 2011-10; Primary Completion 2012-12 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kai Zacharowski, MD, PhD, Principal Investigator — Johann Wolfgang Goethe University Hospital
Locations (1):
- Goethe University Hospital, Frankfurt am Main, Hesse, Germany

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort: Surgical patients from 10 hospitals over a period of 13 months
Period: Overall Study
Arm/Group | Cohort
Started | 10100
Completed | 9103
Not Completed | 997

BASELINE CHARACTERISTICS:
Arm/Group | Cohort
Number analyzed (Participants) | 10100
Age, Customized [Number; unit: years] | NA — Age data not collected.
Sex/Gender, Customized [Number; unit: participants] | NA — Gender data not collected.

OUTCOME MEASURES:

1. Primary Outcome: Number of Different Substitution Solutions Administered
Time Frame: 24h
Population: Surgical patients from 10 hospitals over a period of 13 months
Measure: Number; unit: participants
Groups:
- Crystalloids: crystalloids
- Hydroxyethyl Starch: HES
- Other Colloids: gelatine, albumin,
Arm/Group | Crystalloids | Hydroxyethyl Starch | Other Colloids
Number analyzed (Participants) | 9103 | 9103 | 9103
participants | 7827 | 1055 | 221

ADVERSE EVENTS:
Groups:
- Cohort: Surgical patients
Arm/Group | Cohort
Serious Adverse Events (participants affected / at risk) | 0/10100
Other Adverse Events (participants affected / at risk) | 0/10100

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No